CLINICAL TRIAL: NCT06624917
Title: Assessment of Oncological Safety, Quality of Life, and Environmental Impact of the Green Breast Surgery Protocol
Acronym: BuGs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Gianluca Vanni, Principal Investigator, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BuGS 1.2024
Record Dates: First submitted 2024-09-11; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Female; Breast Cancer; Breast Neoplasms
Keywords: Breast Neoplasm; Environment Related Outcome Measure; Patients' Reported Outcome Measure
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Once enrolled in the study population, patients will be divided prior to admission into the two study groups (Green Breast Surgery Group and Conventional Care Group).
Masking Description: Once enrolled patients were randomized to receive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Breast Surgery (Experimental): Preoperative assessment:
  Counsel patients before admission.
  * Encourage 1 month of no alcohol and smoking before surgery.
  * Recommend weight loss for BMI > 30 with exercise.
  Operative assessment:
  * Admit to Day Surgery Unit.
  * Allow clear liquids until 2 hours before surgery.
  * Give maltodextrin 2 hours prior to surgery.
  * Prescribe antibiotic prophylaxis if needed.
  * Prescribe post-op anti-nausea/vomiting medication.
  * Use Awake Breast Surgery Protocol with Peripheral Nerve Blocks (ESP or PECS1).
  * Follow Intercollage Green Theatre checklist.
  * Post-operative assessment:
  Apply personalized DVT prophylaxis.
  * Allow food and water shortly after surgery.
  * Encourage mobilization a few hours post-surgery.
  * Use telemedicine for first follow-ups and later as needed.
  * Scheduled Time Frame pain (NRS scale) and quality of life (PSQ-18, SF-36, QoL, Breast-Q, TSQ-WT) assessment
  * Check for complications 30 days after surgery.
  Interventions: Procedure: Green Breast Surgery Protocol
- Conventional Surgery (No Intervention): Preoperative assessment:
  Counsel patients before admission.
  * Encourage 1 month of no alcohol and smoking before surgery.
  * Recommend weight loss for BMI > 30 with exercise.
  Operative assessment:
  * Admit to surgical unit according to the surgeon preference
  * Allow clear liquids until 2 hours before surgery.
  * Give maltodextrin 2 hours prior to surgery.
  * Prescribe antibiotic prophylaxis if needed.
  * Prescribe post-op anti-nausea/vomiting medication.
  * Intraoperative management according to Surgeon and Anesthesiologist
  Post-operative assessment:
  * Apply personalized DVT prophylaxis.
  * Allow food and water shortly after surgery.
  * Encourage mobilization according to the intraoperative managment.
  * Use telemedicine for first follow-ups and later as needed.
  * Scheduled Time Frame pain (NRS scale) and quality of life (PSQ-18, SF-36, QoL, Breast-Q, TSQ-WT) assessment
  * Check for complications 30 days after surgery.

INTERVENTIONS:
Procedure: Green Breast Surgery Protocol — A perioperative protocol aiming at reducing environmental impact of surgery, and fast recovery protocol to reduce hospitalization.
  Arms: Green Breast Surgery

SUMMARY:
Breast Cancer (BC) is the primary oncological diagnosis in women, with the annual incidence expected to exceed 3 million new cases by 2040 due to population growth and aging. During the COVID-19 pandemic, novel methods were adopted worldwide to provide continuous patient care, including telehealth, fast-track protocols such as awake surgery in breast cancer.

These innovative techniques allowed for improved access to care, and additionally reduced emissions with environmental impact, better resource utilization, and improved continuity of care, but their impact post-pandemic era has not been investigated.

A current issue is the environmental impact of hospitals, particularly operating rooms, as it has been analysed that 25-30% of hospital waste comes from these areas.

A Breast Green Surgery protocol (BuGS protocol) has been designed to reduce Breast Surgery Impact of care, evaluating for the synergistic effect of different procedure for the first time on classic Clincal Outcome, Patients' Reported Outcome Measure (PROM), and Environment Related Outcome Measure (EROM) in breast cancer surgery.

Main hypothesis is that BuGs protocol will provide a significant reduction in carbon footprint of care (EROM) without impacting clinical outcome and PROMs.

DETAILED DESCRIPTION:
Breast Cancer (BC) is the leading oncological diagnosis in women with an annual incidence of more than 2 million patients diagnosed every year. Because of growing and ageing of population, by 2040 the BC burden is expected to spread over 3 million new cases and 1 million death every year.

Previous studies have shown that utilizing a conservative approach in breast surgery, followed by radiotherapy, leads to higher overall survival compared to radical mastectomy. In such research, survival with conservative surgery appears to be independent of prognostic factors, tumor characteristics, age, and type of therapy. These findings have paved the way for improvements in patient anaesthesiologic experience, transitioning from general anaesthesia to awake surgery, aiming to reduce the impact of post-operative stress on patient recovery.

Conservative surgery allows for a different anaesthesiologic approach, shifting from general anaesthesia to Monitored Anaesthesia Care (MAC). This form of local anaesthesia, accompanied by sedatives and analgesics dosed to allow spontaneous breathing and airway reflexes, promotes quicker post-operative recovery and less psychological impact on the patient compared to general anaesthesia. A comparison between the two techniques was evaluated using the Quality of Recovery-15 (QoR-15) highlighted a higher score with the use of MAC. Moreover, MAC reduces immunomodulation risk in the early postoperative setting, thus reducing potential long-term oncological outcomes on patients, and promoting a novel less immunosuppressive regimen in frail patients. Several studies in oncological patients demonstrated, in these subsets of patients, that the neoplasm may determine a subclinical impairment of immune response with abnormal response toward non-self or neoplastic cells. In fact, in the era of precision oncology, synergistic effects between drugs, general health status (overweight patients), and BC are investigated to underline the beneficial role of general health measures in long-term outcomes.

Additionally, the COVID-19 pandemic represented a practice-changing accelerator in many healthcare services. Many services tried to gather different procedures in a single hospital admission, to reduce the bed occupancy. Among several innovation, a wider application of telehealth demonstrated that many consultations and healthcare services can be effectively delivered via digital platforms. This approach has the potential not only to improve access to care but also to reduce the environmental impact associated with healthcare practices. Telehealth in the context of breast cancer not only offers advantages in terms of accessibility and continuity of care, but also promotes more sustainable healthcare practices, reducing the environmental impact of medical activities.

Aside from mobility for hospital access, the healthcare industry and hospital facilities contribute to environmental pollution. It was estimated in 2013 that 12% of acid rain, 10% of greenhouse gases (GHG), 10% of smog, 1% of ozone gas depletion, and the production of atmospheric carcinogenic and non-carcinogenic toxins derive from healthcare activities within hospitals, with significant implications for public health.

The increase in air pollution and consequently the risk of mortality has led to greater attention to new surgical protocols, which prioritize environmental needs in addition to patient clinical needs due to the resurgence of advanced-stage breast pathology, reduction of operating spaces, and dedicated hospitalization for individual patients. Hospitals and operating rooms represent the primary source of greenhouse gas emissions, with 25-30% of hospital waste being produced by operating rooms.

Due to significant pollutant emissions, hospitals are a major source of environmental impact. In England, the National Health Service (NHS) alone is responsible for emitting 18 million tons of CO2, equivalent to 30% of greenhouse gas emissions from the entire public sector. Therefore, the NHS has initiated reflections and initiatives to make the healthcare sector carbon neutral. Four different intervention phases have been identified, highlighting that reducing CO2 emissions in hospitals, especially in operating rooms, is not simple, mainly due to the current absence of specific guidelines aimed at gas reduction 20. Evaluation parameters, feasibility, and safety have been introduced, expressing percentages at various points from a multicenter study that considers both physicians' and patients' opinions.

A large portion of hospital greenhouse gas emissions comes from the operating room, primarily due to the use of volatile anaesthetics for general anaesthesia. Among these, sevoflurane and desflurane are the main pollutants, from their production in the pharmaceutical sector to their impact on the atmospheric environment, where they persist for several years (1.4 and 21.4, respectively). These compounds act as greenhouse gases, contributing to global warming. Additionally, many volatile anaesthetics contain nitrous oxide (N2O) as a carrier gas, which has a greater impact on global warming when mixed with ambient air 23. This complex process, from pharmaceutical production to the atmosphere, represents a significant source of greenhouse gases originating from the hospital setting.

It has been shown that reducing the use of anaesthetics, especially the volatile ones, in surgery is possible, particularly highlighted by Wide-Awake Local Anaesthesia No-Tourniquet (WALANT) surgery performed for small ambulatory hand operations. Patient satisfaction and better resource allocation are the most significant post-operative benefits of WALANT. Studies have reported that 94% of patients would choose WALANT again in the future. Patients experience reduced post-operative pain compared to previous surgeries with tourniquet sedation. WALANT promotes better communication between the patient and the surgical team, enhancing understanding, compliance, and prevention of post-operative injuries. It reduces time spent in the post-operative phase, resulting in decreased costs for both the facility and the patient.

Reducing surgical impact has been a recent theme in general surgery. Since the 2000s, numerous authors have begun outlining the so-called Enhanced Recovery After Surgery (ERAS) protocols in general surgery, especially in colorectal surgery 26,27. This multidisciplinary protocol aims to improve outcomes after surgery, articulating into four phases to ensure better control and greater adherence to the correct course: pre-hospitalization, pre-operative, intra-operative, and post-operative. Regarding colorectal surgery, ERAS programs have shown improvements in post-operative hospitalization times, mortality, and consequently increased long-term survival. Specifically, in patients with ≥70% adherence to the ERAS protocol, the 5-year specific cancer death risk decreased by 42%.

From the results of studies conducted using ERAS and WALANT approaches, as well as telehealth assistance, it has emerged that their protocols can be effectively applied in breast surgery. In fact, in the recent years, awake surgery plus locoregional anesthetic regimen emerged as novel approach to accelerate postoperative recovery and minimize postoperative complication. Consequently, our group is committed to implementing such studies and evaluating the results obtained.

The ERAS protocol can also be applied in the field of breast surgery, which, together with telehealth in the peri-operative and post-operative pathways, lays the groundwork for the Green Breast Surgery research project. This pathway is dedicated to patients undergoing conservative surgical treatment for breast pathology and is based on the analysis of clinical outcomes, quality of life, as well as social, environmental, and economic effects in the application of this telehealth protocol in clinical practice.

Limiting the resources applied in operating rooms allows for a greater number of patients to undergo surgical procedures, particularly in the field of senology. The reason why the Breast Unit is a good candidate for this type of protocol lies in the possibility of operating on the patient while awake, without the need for general anaesthesia, due to the simplicity of the surgical procedure itself.

A recent study has highlighted how climate change exacerbates health problems and creates new ones, particularly in low-income countries. Among the effects of climate change, increasing temperatures lead to a higher frequency of surgical site infections by up to 39%, while air pollution causes prolonged hospital stays and increased costs. A protocol has been implemented with five different aspects of the surgical setting that can be improved, ranging from the use of non-volatile anaesthetics to modifying some behaviors of operating room staff such as reducing the use of syringes, turning off lights when the operating room is not in use, and implementing telehealth instead of outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for Breast Conserving Treatment
* ASA score I-II
* Availability to Telehealth assessment in the postoperative period

Exclusion Criteria:

* Drug addiction
* contraindication for locoregional ultrasound-guided procedure (e.g., local infection, allergy to LA)
* chronic pain under treatment
* pregnancy
* No follow-up planned in our facility

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
24 h Post-operative pain at rest | 24 hours after surgery
  Postoperative Pain at rest with Numeric Pain Rating Scale NPRS (0-10)
24 h Post-operative dynamic pain | 24 hours after surgery
  Postoperative dynamic Pain with Numeric Pain Rating Scale NPRS (0-10)

SECONDARY OUTCOMES:
Number of hospital admissions after surgery | 30 days after surgery
  Number of hospital admissions after surgery
Assessment Telehealth implementation | 30 days after surgery
  Assessment Telehealth implementation with Telemedicine Satisfaction Questionnaire (TSQ)
Patients' reported outcome measures | 30 days after surgery
  Patients' reported outcome measures with Short-Form Patient Satisfaction Questionnaire (PSQ-18)
Patients' reported outcome measures | 30 days after surgery
  Patients' reported outcome measures with The Short Form (36) Health Survey (SF-36)
Patients' reported outcome measures | 30 days after surgery
  Patients' reported outcome measures with BREAST-Q Breast-Conserving Therapy Module
48 hours Post-operative pain at rest | 30 days hours after surgery
  Postoperative Pain at rest with Numeric Pain Rating Scale NPRS (0-10)
48 hours Post-operative dynamic pain | 30 days hours after surgery
  Postoperative dynamic pain with Numeric Pain Rating Scale NPRS (0-10)
30 days Post-operative pain at rest | 30 days after surgery
  Postoperative Pain at rest with Numeric Pain Rating Scale NPRS (0-10)
30 days Post-operative dynamic pain | 30 days after surgery
  Postoperative dynamic pain with Numeric Pain Rating Scale NPRS (0-10)
Carbon footprint of surgery room | Time of surgery
  Evaluation of waste produced in the surgical room (reciclable waste, infected waste, non infected waste)
Hospitalization | Time of Surgery
  Days of hospitalization
30 Days surgical complication | 1 months
  30 Days surgical complication evaluated with Clavien Dindò modified classification for breast cancer

OTHER OUTCOMES:
Carbon footprint of private patient transport to the hospital | 30 days after surgery
  Carbon footprint of private patient transport

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Vanni, PhD, Principal Investigator — University of Rome Tor Vergata; Oreste Claudio Buonomo, Full Prof, Study Chair — University of Rome Tor Vergata
Locations (1):
- Università degli Studi di Roma Tor Vergata, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Materazzo M., Facchini A., Garozzo D., Buonomo C., Pellicciaro M., Vanni G. Maintaining good practice in breast cancer management and reducing the carbon footprint of care: study protocol and preliminary results WCRJ 2022; 9: e2438 DOI: 10.32113/wcrj_202211_2438
- [Background] Vanni G, Caiazza G, Materazzo M, Storti G, Pellicciaro M, Buonomo C, Natoli S, Fabbi E, Dauri M. Erector Spinae Plane Block Versus Serratus Plane Block in Breast Conserving Surgery: Alpha Randomized Controlled Trial. Anticancer Res. 2021 Nov;41(11):5667-5676. doi: 10.21873/anticanres.15383. PMID 34732440
- [Background] Vanni G, Materazzo M, Pellicciaro M, Marino D, Buonomo OC. From Patient Reported Outcome Measure (PROM) to Environment Related Outcome Measure (EROM): Towards "Green Breast Surgery". In Vivo. 2023 Jul-Aug;37(4):1867-1872. doi: 10.21873/invivo.13278. PMID 37369495